CLINICAL TRIAL: NCT03837041
Title: Evaluate the Proprioception in Patients with Total Knee Arthroplasty
Brief Title: Evaluation of Proprioception
Acronym: PROPRIO_TPG
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Istituto Ortopedico Rizzoli (Other)
Collaborators: University of Bologna (Other)
Responsible Party: Principal Investigator, Stefano Zaffagnini, Full Professor and Head of department, Istituto Ortopedico Rizzoli
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: PROPRIO_TPG
Record Dates: First submitted 2019-02-07; First posted 2019-02-11 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2023-05

CONDITIONS: Proprioceptive Disorders
Keywords: total knee arthroplasty; Proprioception; osteoarthritis
MeSH Terms: conditions — Somatosensory Disorders; Osteoarthritis

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Reconditioning Proprioception group (Active Comparator): Training Proprioception 1 hour for 2 day a week
  Interventions: Other: Reconditioning Proprioception
- Control group (No Intervention)

INTERVENTIONS:
Other: Reconditioning Proprioception — Proprioceptive training using Delos Postural Proprioceptive System
  Arms: Reconditioning Proprioception group

SUMMARY:
The osteoarthritis (OA) is a chronic and degenerative disease which brings articular cartilage degeneration. As a consequence, balance and proprioception could be dangerously reduced after total knee arthroplasty.

Several studies demonstrated the correlation between OA, proprioception reduction and increased risk of falling. The aim of this study is to evaluate the proprioception improvement in patients with total knee arthroplasty.

ELIGIBILITY:
Inclusion Criteria are patients with ASA: 1, 2 or 3; patients who have given their informed written consent to participate in the study; patients live in Bologna and neighboring areas.

Exclusion Criteria are patients with previous osteotomy of the lower limbs; patients with post-traumatic arthrosis; patients with severe preoperative valgus deformity (Hip Knee Ankle angle> 10 °); patients with BMI> 40 kg / m2; patients with rheumatoid arthritis; patients with chronic inflammatory joint diseases; patients with walking diseases (amputations, neuro-muscular diseases, polio, hip dysplasias); patients with Severe arthrosis of the ankle (Kellgren-Lawrence> 3); patients with Severe coxarthrosis (Kellgren-Lawrence> 3); patients with severe postural instability; patients with cognitive impairments, patients with concomitant neurological diseases

Ages: 45 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 71 (Actual)
Dates: Start 2017-03-01 (Actual); Primary Completion 2021-07-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Improvement of a proprioception | 24 months
  Stability Index (SI) in percentage the maximum is 100%

SECONDARY OUTCOMES:
Evaluation of performance in lower limb questionnaire | 24 months
  Short Physical Performance Battery - SPPB The score range from 0 (wost performance) to 12 (best performance)
KSS Score | 24 months
  The score range from 0 to 100 with lower scores being indicative of worse knee conditions and higher scores being indicative of better knee conditions
Clinical score | 24 months
  Western Ontario and McMaster Universities Osteoarthritis Index the WOMAC evaluates 3 dimensions: pain, stiffness, and physical function with 5, 2, and 17 questions, respectively. The Likert version of the WOMAC is rated on an ordinal scale of 0 to 4, with lower scores indicating lower levels of symptoms or physical disability.

CONTACTS AND LOCATIONS:
Locations (1):
- Istituto Ortopedico Rizzoli, Bologna, Bologna, Italy

IPD SHARING:
Plan to Share IPD: Undecided